CLINICAL TRIAL: NCT00802646
Title: Randomized, Double-Blind, Placebo-Controlled Study of Effects of Combined Spinal Epidural Analgesia on Intrapartum Fever.
Brief Title: The Effects of Combined Spinal Epidurals on Fever During Labor of First-Time Mothers
Acronym: CSE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study moved to alternate site
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2008.; 2008.
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Vaginal Delivery
Keywords: first-time mother; epidural request; vaginal childbirth
MeSH Terms: interventions — Sodium Chloride; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): When it is time for the epidural catheter, the mother will receive 2.5 mcg fentanyl spinally and then a bag of preservative-free normal saline will be administered through the epidural pump. When additional pain medication is requested, the mother will receive a known combined spinal epidural solution.
  Interventions: Drug: saline
- 2 (Active Comparator): When it is time for the epidural catheter, the mother will receive 2.5 mcg fentanyl spinally and then a bag of combined spinal epidural anesthetic through the epidural pump. When additional pain medication is requested, the mother will receive a known combined spinal epidural solution.
  Interventions: Drug: fentanyl/bupivacaine/epinephrine

INTERVENTIONS:
Drug: saline — intrathecal preservative free normal saline, 8ml/hour, beginning after intrathecal sufentanyl until additional pain medication is requested
  Other Names: placebo
  Arms: 1
Drug: fentanyl/bupivacaine/epinephrine — intrathecal 0.125% fentanyl/bupivacaine/epinephrine, 8ml/hour, beginning after intrathecal sufentanyl until additional pain medication is requested The mother will then receive a new bag of fentanyl/bupivacaine/epinephrine.
  Other Names: combined spinal epidural
  Arms: 2

SUMMARY:
The purpose of this study is to determine if the epidural of local anesthetics has an effect on fever that may occur in first time mothers during labor.

DETAILED DESCRIPTION:
Intrapartum fever (fever during labor) is a real and potentially devastating problem. Infants delivered at term who have been exposed to the mother having a fever during labor have a >9 fold increased risk of cerebral palsy. Studies have also shown an increased risk of neonatal encephalopathy associated with fever during labor. Maternal fever in the absence of infection is associated with a 4 fold increased risk of neonatal hypoxic encephalopathy and 3.4 fold increased risk of unexplained neonatal seizures.

The likely role of inflammatory mediators in the process of maternal fever (temperature >100.4), regardless of etiology, makes it important to further investigational studies in an effort to discover the etiology of intrapartum fever associated with epidural analgesia. If an inflammatory trigger (i.e., the injection of epidural local anesthetics) can be identified or delayed, then the risks of maternal hyperthermia can be minimized and/ or eliminated.

The greatest risk of fever with epidural labor analgesia is seen in women having their first child. This is the same population associated with prolonged labor. Although intrapartum fever has a very low incidence overall, 11-33% of first-time mothers will eventually develop fever >100.4 during epidural analgesia. Although the degree of rise in temperature occurs very slowly, it has been shown to be significant enough to cause increased neonatal sepsis workup and antibiotic coverage for both the mother and the neonate.

ELIGIBILITY:
Inclusion Criteria:

* having first child (nulliparous)
* term pregnancy (> 37 weeks)
* vertex presentation
* singleton gestation
* ability to provide informed consent
* request for analgesia for labor pain

Exclusion Criteria:

* birth of second or more child (multiparous)
* preterm pregnancy (< 37 weeks)
* presentation other than vertex (ie. breech, transverse)
* diabetic
* admit temperature > 99.5
* active drug/alcohol dependence
* active genital herpes infection
* allergy to anesthetics used

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
temperature of mother | time of delivery

SECONDARY OUTCOMES:
neonatal APGAR, temperature and cord blood gas | time of birth

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Russo, M.D., Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Lieberman E, Eichenwald E, Mathur G, Richardson D, Heffner L, Cohen A. Intrapartum fever and unexplained seizures in term infants. Pediatrics. 2000 Nov;106(5):983-8. doi: 10.1542/peds.106.5.983. PMID 11061764
- [Background] Lieberman E, Lang JM, Frigoletto F Jr, Richardson DK, Ringer SA, Cohen A. Epidural analgesia, intrapartum fever, and neonatal sepsis evaluation. Pediatrics. 1997 Mar;99(3):415-9. doi: 10.1542/peds.99.3.415. PMID 9041298
- [Background] Yancey MK, Zhang J, Schwarz J, Dietrich CS 3rd, Klebanoff M. Labor epidural analgesia and intrapartum maternal hyperthermia. Obstet Gynecol. 2001 Nov;98(5 Pt 1):763-70. doi: 10.1016/s0029-7844(01)01537-x. PMID 11704166
- [Background] Fusi L, Steer PJ, Maresh MJ, Beard RW. Maternal pyrexia associated with the use of epidural analgesia in labour. Lancet. 1989 Jun 3;1(8649):1250-2. doi: 10.1016/s0140-6736(89)92341-6. PMID 2566791
- [Background] Leighton BL, Halpern SH. The effects of epidural analgesia on labor, maternal, and neonatal outcomes: a systematic review. Am J Obstet Gynecol. 2002 May;186(5 Suppl Nature):S69-77. doi: 10.1067/mob.2002.121813. PMID 12011873
- [Background] Dashe JS, Rogers BB, McIntire DD, Leveno KJ. Epidural analgesia and intrapartum fever: placental findings. Obstet Gynecol. 1999 Mar;93(3):341-4. doi: 10.1016/s0029-7844(98)00415-3. PMID 10074975
- [Background] Kaul B, Vallejo M, Ramanathan S, Mandell G. Epidural labor analgesia and neonatal sepsis evaluation rate: a quality improvement study. Anesth Analg. 2001 Oct;93(4):986-90. doi: 10.1097/00000539-200110000-00038. PMID 11574370
- [Background] Goodlin RC, Chapin JW. Determinants of maternal temperature during labor. Am J Obstet Gynecol. 1982 May 1;143(1):97-103. doi: 10.1016/0002-9378(82)90689-5. PMID 7081319
- [Background] Gleeson NC, Nolan KM, Ford MR. Temperature, labour, and epidural analgesia. Lancet. 1989 Oct 7;2(8667):861-2. doi: 10.1016/s0140-6736(89)93020-1. No abstract available. PMID 2571778
- [Result] Grether JK, Nelson KB. Maternal infection and cerebral palsy in infants of normal birth weight. JAMA. 1997 Jul 16;278(3):207-11. PMID 9218666
- [Result] Impey L, Greenwood C, MacQuillan K, Reynolds M, Sheil O. Fever in labour and neonatal encephalopathy: a prospective cohort study. BJOG. 2001 Jun;108(6):594-7. doi: 10.1111/j.1471-0528.2001.00145.x. PMID 11426893
- [Result] Sharma SK, Alexander JM, Messick G, Bloom SL, McIntire DD, Wiley J, Leveno KJ. Cesarean delivery: a randomized trial of epidural analgesia versus intravenous meperidine analgesia during labor in nulliparous women. Anesthesiology. 2002 Mar;96(3):546-51. doi: 10.1097/00000542-200203000-00007. PMID 11873026
- [Result] Ramin SM, Gambling DR, Lucas MJ, Sharma SK, Sidawi JE, Leveno KJ. Randomized trial of epidural versus intravenous analgesia during labor. Obstet Gynecol. 1995 Nov;86(5):783-9. doi: 10.1016/0029-7844(95)00269-w. PMID 7566849
- [Result] Goetzl L, Cohen A, Frigoletto F Jr, Lang JM, Lieberman E. Maternal epidural analgesia and rates of maternal antibiotic treatment in a low-risk nulliparous population. J Perinatol. 2003 Sep;23(6):457-61. doi: 10.1038/sj.jp.7210967. PMID 13679931
- [Result] Goetzl L, Rivers J, Evans T, Citron DR, Richardson BE, Lieberman E, Suresh MS. Prophylactic acetaminophen does not prevent epidural fever in nulliparous women: a double-blind placebo-controlled trial. J Perinatol. 2004 Aug;24(8):471-5. doi: 10.1038/sj.jp.7211128. PMID 15141263
- [Result] Goetzl L, Zighelboim I, Badell M, Rivers J, Mastrangelo MA, Tweardy D, Suresh MS. Maternal corticosteroids to prevent intrauterine exposure to hyperthermia and inflammation: a randomized, double-blind, placebo-controlled trial. Am J Obstet Gynecol. 2006 Oct;195(4):1031-7. doi: 10.1016/j.ajog.2006.06.012. Epub 2006 Jul 26. PMID 16875647
- [Result] Banerjee S, Cashman P, Yentis SM, Steer PJ. Maternal temperature monitoring during labor: concordance and variability among monitoring sites. Obstet Gynecol. 2004 Feb;103(2):287-93. doi: 10.1097/01.AOG.0000100155.85379.88. PMID 14754697
- [Result] Arkoosh VA, Palmer CM, Yun EM, Sharma SK, Bates JN, Wissler RN, Buxbaum JL, Nogami WM, Gracely EJ. A randomized, double-masked, multicenter comparison of the safety of continuous intrathecal labor analgesia using a 28-gauge catheter versus continuous epidural labor analgesia. Anesthesiology. 2008 Feb;108(2):286-98. doi: 10.1097/01.anes.0000299429.52105.e5. PMID 18212574